CLINICAL TRIAL: NCT02499926
Title: Determination of Lysine Oxidation in Response to Arginine Supplementation in Adult Men Using in Vivo Stable Isotope Techniques
Brief Title: Lysine Oxidation in Response to Arginine Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Rajavel Elango, PhD, Assistant Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H15-01151
Record Dates: First submitted 2015-07-14; First posted 2015-07-16 (Estimated); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Physiologically Healthy Adult Male Participants
MeSH Terms: interventions — Arginine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dietary supplement: Arginine (Experimental): Graded arginine excess intake
  Interventions: Dietary Supplement: Arginine

INTERVENTIONS:
Dietary Supplement: Arginine — Graded arginine excess intake will start at 50mg/kg/d on study day 1 followed by 100 mg/kg/d on study day 2 till the level reaches 300mg/kg/d on study day 6.
  Consisting of oral consumption of eight hourly experimental meals per study day - Includes 4 tracer free experimental meals containing a mixture of free amino acids, calories from a flavored liquid and protein free cookies and 4- labeled amino acid experimental meals.

SUMMARY:
This research study is investigating if consuming more of one amino acid (arginine) influences the digestion and absorption of another amino acid (lysine) due to competition in digestion, in a healthy adult population.

DETAILED DESCRIPTION:
Background:

Protein is made up of building blocks called amino acids. Some amino acids, including Lysine, cannot be made in the body and must be obtained from diet, and these are called essential amino acids.

Pyridoxine dependent deficiency (PDE) is a rare condition caused by the body's inability to properly breakdown lysine. This is due to a missing enzyme, α- aminoadipic semi-aldehyde dehydrogenase (α-AASAD) also known as antiquitin (ATQ), involved in lysine breakdown. When the enzyme is missing and/or not functioning properly, it increases the level of byproducts of lysine breakdown that may result in seizures babies and young children and affect brain development. As with many other similar conditions, a low lysine diet may be helpful for some patients, but can pose a significant burden on the patient and the families.

More recently, animal experiments have shown that the body's ability to absorb lysine from the diet can be altered by adding more of another "competitive" amino acid, in this case, arginine. This is because lysine and arginine share the same transport system in the body.

Therefore, the current study is designed to describe the application of 13C-lysine to explore the changes in lysine breakdown caused by varying (graded) amounts of arginine supplementation in young adult male participants.

Study design:

Two adult male subjects aged 19-50 y will be recruited to participate in 6 graded doses of arginine intakes, in addition to a test diet which will provide the lysine at normal intake of 110mg/kg/d. Lysine intake levels, will be determined based on subject age and body weight and will remain constant for the entire study period. The recommended dietary protein intake (DRI) will be maintained throughout the study.

A thorough pre-study assessment will be performed and all subjects will be screened by questionnaire for chronic diseases, physical activity and dietary habits. Lean body mass or skeletal muscle mass (Bioelectrical impedance Analysis) will be measured. Subjects will be ensured to be free of chronic diseases.

Arginine Test Intakes:

Graded arginine excess intake will start at 50mg/kg/d on study day 1 followed by 100 mg/kg/d on study day 2 till the level reaches 300mg/kg/d on study day 6.

The arginine test intakes will be provided in the form of protein shakes containing a stable isotope, and then oxidation of this isotope will be measured to determine whether arginine that will competitively inhibit lysine uptake.

To measure how the the body responds to the test diet we will collect seven breath samples, two urine samples and one blood sample during each study day.

ELIGIBILITY:
Inclusion Criteria:

* You are 19 to 50 years-of-age
* Male
* Classified as normal body weight and BMI (18.5-25 kg/m2)
* Free of any concurrent illness (cold, flu, vomiting etc.)
* Not be claustrophobic (we will place a clear hood, which can easily be removed, over your head for approximately 20 min to measure your energy expenditure).
* Not be enrolled in any other research studies (as this may affect our study results)

Exclusion Criteria:

You are not in good health or have a metabolic, neurological, genetic, or immune disorder, including diabetes and hypertension

* You are classified as underweight (<18.5 kg/m2), overweight (25-30 kg/m2), or obese (>30 kg/m2) using the BMI classification
* You are allergic to milk, eggs and egg protein
* You are claustrophobic (we will place a clear hood, which can easily be removed, over your head for approximately 20 min to measure your energy expenditure)
* You are currently enrolled in other research studies (as this may affect our study results)

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2015-07; Primary Completion 2017-12 (Actual); Study Completion 2024-01-12 (Actual)

PRIMARY OUTCOMES:
13CO2 production | 8 hours (1 study day)
  Urine, plasma and breath samples will be collected during the study to measure the rate of oxidation of tracer with graded intake of arginine

CONTACTS AND LOCATIONS:
Overall Officials: Rajavel Elango, PhD, Principal Investigator — University of British Columbia
Locations (1):
- BC Children;s Hospital Research Institute, University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No